CLINICAL TRIAL: NCT03793673
Title: CoYoT1 to California - Telemedicine to Engage Young Adults With Diabetes
Brief Title: CoYoT1 to California
Acronym: CTC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Los Angeles (Other)
Collaborators: University of Southern California (Other); Rutgers University (Other)
Responsible Party: Principal Investigator, jennifer raymond, MD, MCR, Associate Professor of Clinical Pediatrics, Clinical Director of Diabetes Center for Endocrinology, Diabetes, and Metabolism, Vice Chair of the Executive Telehealth Committee, Children's Hospital Los Angeles
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Other
Other Study IDs: CHLA-18-00488
Record Dates: First submitted 2018-11-23; First posted 2019-01-04 (Actual); Last update posted 2023-03-15 (Actual); Status verified 2023-03

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: Adolescents and Young Adults(AYA)
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Standard Care: Standard appointments (Other): Usual in-person medical appointments. See previous detailed description.
  COVID-19 Update: Current clinic appointments consist of telehealth appointments only. Any additional community and CHLA based educational and support events will be following COVID-19 guidelines.
  Interventions: Other: Standard Care
- Standard Care: Telehealth appointments (Other): Telehealth - with provider and/or team. See previous detailed description.
  Interventions: Other: Standard Care
- CoYoT1 Care: Standard Appointment (Other): In-person - medical appointments with provider and/or team. See previous detailed description.
  COVID-19 Update: Current clinic appointments consist of telehealth appointments only. Any additional community and CHLA based educational and support events will be following COVID-19 guidelines.
  Interventions: Behavioral: CoYoT1 Care
- CoYoT1 Care: Telehealth appointments (Other): Telehealth - with provider and/or team. See previous detailed description.
  Interventions: Behavioral: CoYoT1 Care

INTERVENTIONS:
Behavioral: CoYoT1 Care — Selected providers will be trained in the CoYoT1 Care protocol for completing medical appointments (both telehealth/standard appointments). There are three key components: (1) Shared decision making: Providers and YA will mutually agree on priorities for each medical visit using a shared decision making tool completed by both the provider and patient. (2) Autonomy supportive care: Providers will be trained in communication strategies, such as motivational interviewing, designed to support YA autonomy and intrinsic motivation. YA will also direct extent of eligible family involvement. (3) Goal setting and action planning: Providers will be trained to coach YA in setting SMART goals, developing action plans, and establishing a plan for follow-up between visits as appropriate.
  Arms: CoYoT1 Care: Standard Appointment; CoYoT1 Care: Telehealth appointments
Other: Standard Care — Providers selected for the Standard Care group will complete medical appointments in their usual manner, without specific training or guidelines regarding how to deliver care.
  NOTE: Per COVID-19 hospital policies, current clinic appointments consist of telehealth appointments.
  Arms: Standard Care: Standard appointments; Standard Care: Telehealth appointments

SUMMARY:
CoYoT1 to California (CTC) was initiated to develop a patient-centered, home telehealth care model for young adults (YA) ages 16-25 with T1D. It is a 2x2 factorial design, 15-month intervention. Eighty participants will be randomized to Standard Care or CoYoT1 Care, which is delivered by telehealth or in-person. CoYoT1 Care is a patient-centered care model that consists of three major components: shared decision making (patient and provider agree upon priorities for the medical visit), autonomy and supportive care (provider training in communication strategies such as motivational interviewing), and goal setting and action planning (provider training to coach YA in setting SMART goals, developing action plans, and designing follow up plans). Additionally, didactic expert-led sessions (Standard Care) or peer-led, YA-driven group sessions (CoYoT1 Care) are included. At the end of the study, a focus group will be completed to assist in determining which features YA felt were critical to their success from the telehealth intervention, group components, and provider behaviors.

***COVID-19 Update: Due to current hospital and clinical policy adaptation for COVID-19, all participants who were randomized into in-person appointments will now receive care via Telehealth. Telehealth has been implemented hospital-wide and will be the temporary delivery of care method during this pandemic. Participants have been notified of this change and given instruction on how to participate in a Telehealth appointment.

DETAILED DESCRIPTION:
1. Standard Care - Standard (in -person) appointments

   * Usual medical appointments.
   * Opportunity to participate in available community and CHLA based educational and support events.
   * Complete online assessments/questionnaires.
   * Invitation to a 2 hour audio-recorded discussion at the end of the study

     * COVID-19 Update: Current clinic appointments consist of telehealth appointments only. Any additional community and CHLA based educational and support events will be following COVID-19 guidelines.
2. Standard Care - Telehealth appointments

   * Telehealth - with provider and/or team. Online video appointments every 3 months, upload diabetes data to Tidepool, and do routine blood work at a facility near you
   * Opportunity to participate in available community and CHLA based educational and support events
   * Complete online assessments/questionnaires
   * Invitation to a 2 hour audio-recorded discussion at the end of the study

     * COVID-19 Update: Any community and CHLA based educational and support events will be following COVID-19 guidelines. If in-person routine bloodwork is not feasible, HbA1c kits will be provided to participants.
3. CoYoT1 Care - Standard Appointment

   * In-person - medical appointments with provider and/or team
   * Opportunity to participate in 30-60 minute online peer-led diabetes group discussions
   * Complete online assessments/questionnaires
   * Invitation to a 2 hour audio-recorded discussion at the end of the study

     * COVID-19 Update: Current clinic appointments consist of telehealth appointments only.
4. CoYoT1 Care - Telehealth appointments

   * Telehealth - with provider and/or team. Online video appointment every 3 months, upload your diabetes data to Tidepool, and do routine blood work at a facility near you
   * Opportunity to participate in 30-60 minute online peer-led diabetes group discussions
   * Complete online assessments/questionnaires
   * Invitation to a 2 hour audio-recorded discussion at the end of the study

     * COVID-19 Update: If in-person routine bloodwork is not feasible, HbA1c kits will be provided to participants.

ELIGIBILITY:
Inclusion Criteria:

* Any patient aged 16-25 years of age on their date of recruitment who has had T1D for at least 6 months.
* Receiving or pending care at CHLA
* Has California Children's Services (CCS), self-pay, and/or private insurance (excluding United and Healthnet insurance)
* Does not plan to transfer out of CHLA within the next year

Exclusion Criteria:

* Any patient with severe behavioral or developmental disabilities
* Severe psychological diagnoses that would make group participation difficult
* Pregnancy
* Non-English speaking patients and families
* Has United or Healthnet private insurance
* Literacy or cognitive issues that preclude the use of the Internet

Ages: 16 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 82 (Actual)
Dates: Start 2019-01-20 (Actual); Primary Completion 2022-07-28 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Number of participants with completed appointments in telemedicine cohort | 12 months
  Electronic Medical Record (EMR) Abstraction - number of appointments; multiple choice and open ended
Number of participants with completed appointments in telemedicine cohort | 12 months
  Patient online attendance as assessed using an online patient experience questionnaire - Polar Questions; Yes or no response questions related to patient's online appointment (i.e., did you have an online appointment? Did you attend your appointment?)
Number of participants with completed medical appointments in standard care cohort | 12 months
  In-person patient appointment attendance assessed using an online patient experience questionnaire. Polar questions; Yes or No response questions related to patient's in-person appointment (i.e., did you have an in-person appointment? Did you attend your in-person appointment?
Patient and Provider Satisfaction as assessed using the Health Care Climate questionnaire | 12 months
  : Likert scale "Very dissatisfied" is 1, "Dissatisfied" is 2, "Neutral" is 3, "Satisfied" is 4, and "Very Satisfied" is 5. Higher scores indicate more satisfaction, lower scores indicate low satisfaction
Provider Experience as assessed using the CAHPS survey | 12 months
  Cultural Competence Consumer Assessment of Healthcare Providers and Systems (CAHPS) - likert Scale; range 0-10, low range indicates low trust and high values indicate trust.
Patient Satisfaction with appointment type as assessed using the Updated CoYoT1 Satisfaction Questionnaire | [Time Frame: For each visit (until the end of study) - 12 months]
  Likert scale; "Strongly disagree" is 1, "Somewhat disagree" is 2, "Neutral" is 3, "Somewhat Agree" is 4, and "Strongly Agree" is 5. Scores are summed and the average is taken; higher scores is more self-efficacy
Provider Satisfaction as assessed using the Satisfaction Provider survey | 12 months
  Telehealth Utilization satisfaction as assessed using a telehealth satisfaction questionnaire. Likert scale; range 1-5, low values indicate low satisfaction and higher values indicate high satisfaction. Polar: Yes or No response questions, "Would you use telehealth again?" Open ended; patient comments about experience.
Patient Experience | 12 months
  Patient Experience Measures Consumer Assessment of Healthcare Providers and Systems (CAHPS) - likert Scale; range 0-10; lower range represents low rating, higher ranges indicate higher rating
Social Determinants of Health Tool | At 0 (baseline)
  Social determinants of health as assessed using a social and environmental factors questionnaire. Polar; Yes or No questions about food insecurity and transportation, "did you worry that your food would run out before you got money to buy more?" "have you or your family ever been unable to go to the doctor because of distance or transportation?"

SECONDARY OUTCOMES:
Costs to Patients | 12 months
  Transportation cost to patient as assessed using a Transportation Questionnaire. Multiple choice questions about mode of transportation used to get to appointment, "driving own vehicle," "riding public transit," "ride with family member or friend." Open ended to assess cost of parking, bus fare.
Costs to Patients | 12 months
  Number of patients with need for a technology device (cellphone) as assessed using a Device Assessment questionnaire. Polar; Yes or No question about access to personal device patient has for online appointment, "do you have a personal device to access the internet?." Multiple choice questions about device; "Mobile phone," "Laptop," "Tablet," "Ethernet," "Wi-Fi."
Costs to Patients | 12 months
  Diabetes visit expenses questions - polar questions, multiple choice, and open-ended
Cost to Instituition | 12 months
  Cost to Institution as assessed by Patient Health Utilization questionnaire. Polar; Yes or No questions about health service usage in the last three months, "have you had to be admitted to the hospital?" Open-ended question about number of time health services were used, "how many times were you admitted to the hospital for reasons related to diabetes?"
Cost to Instituition | 12 months
  Cost to Institution as assessed using the Online Appointment questionnaire. Polar; Yes or No questions about attendance to online appointment. "Did you attend your online appointment?" "What types of providers did you see?" Open-ended questions asking about time, "how long did it take?"
Cost to Instituition | 12 months
  Cost to Institution as assessed using the In-Person Appointment questionnaire. Polar; Yes or No questionnaire about appointment attendance; "did you attend an in-person appointment?" "How long was your in-person appointment?" Open-ended questions about time, "how long did it take?"
Cost to Instituition | 12 months
  Cost to Institution as assessed using the Clinic Cost, Preparation, and Delivery for Providers and Staff questionnaire. Multiple choice questions about person (Doctor, Nurse and Social Worker) and appointment type provided to patient
Cost to Instituition | 12 months
  Cost to Institution as assessed using Team Costs of Provider and Staff Training questionnaire. Multiple choice questions used to identify person being trained, "Doctor," "Nurse Practitioner," "Social Worker." Polar; Yes or No questions about provider and staff training for telehealth appointment; training on, "camera and mic," "loading Webex platform."
Glycemic Control at Baseline | HbA1c for the last 12 months
  Lab Results: Electronic Medical Record Hemoglobin A1c (HbA1c) %
Glycemic Control Progression | For each visit (until the end of study) - 12 months
  Lab Results: Electronic Medical Record Hemoglobin A1c (HbA1c) %
Cost to Payor | 12 months (monthly)
  Cost to Payor as assessed using Health Care Utilization Online questionnaire. Polar; Yes and No questions about patient use of health services, "In the last 3 months, has 911 been called because of your diabetes?" Open-ended questions about rate of health service use, "how many times was 911 called?"
Cost to Payor | 12 months
  Cost to payor as assessed using Clinic Cost, Preparation, and Delivery questionnaire for Providers or Staff. Open ended questions about length of training and technology used, along with any comments about appointment delivery.
Cost to Payor | 12 months
  Cost to payor as assessed using the Team Costs of Provider or Staff questionnaire. Open ended question asking about length of training and training required on "billing process," "data collection process," "camera and mic."
Cost to Payor as as assessed using the Team Costs- YA | 12 months
  Multiple Choice and fill-in. Questions about time spent training young adults and training required on "Agenda setting", "Camera and Mic", "Loading Webex platform".

OTHER OUTCOMES:
Self-care, mobility, and anxiety and depression as assessed using the EuroQOL five dimensions five levels questionnaire (EQ-5D-5L) questionnaire. | At 0 (baseline) and 12 months (after visit 4)
  Likert scale; used to measure respondents' endorsement of particular statements. Descriptive system top answer is 1 and last answer is 5. Missing items will be coded as 9. Online software used to score.
Depressive symptoms assessed using the Center of Epidemiologic Studies Scale (CES-D) | At 0 (baseline) and 12 months (after visit 4)
  "Rarely or none of the time (less than 1 day)" is 0, "Some or a little of the time (1-2 days)" is 1, "Occasionally or a moderate amount of time" is 2, "Most or all of the time (5-7 days)" is 3. The scoring of positive items is reversed. Possible range of scores is zero to 60, with the higher scores indicating the presence of more symptomatology.
Patient health-related quality of life as assessed using the Your Health and Well-being Short-Form 12 item Version 2 (SF12V2) measure | At 0 (baseline) and 12 months (after visit 4)
  Likert scale; "Excellent" is 1, "Very good" is 2, "Good" is 3, "Fair" is 4, and "Poor" is 5. An algorithm is used to generate the physical and mental health composite scores for comparison (a confirmatory factor analyses).Items are scored so that a higher score indicates a better health state.
Dimensions of distress (e.g., emotional burden, regimen distress, interpersonal distress and physician distress) as assessed using the Diabetes Distress Scale (DDS) | At 0 (baseline) and 12 months (after visit 4)
  Likert scale; "Not a problem" is 1, "A slight problem" is 2, "A moderate problem" is 3, "Somewhat serious problem" is 4, "A Serious Problem" is 5, and "A very serious problem" is 6. There are 4 subscales that address the dimensions of distress and to score, the appropriate item(s) are summed and divided by appropriate number. A mean item score of 3 or higher is considered moderate distress.
  burden, regimen distress, interpersonal distress and physician distress; likert scale
Assessment of Diabetes-Related Psychosocial Self-Efficacy | At 0 (baseline) and 12 months (after visit 4)
  Diabetes-related psychosocial self-efficacy as assessed using the Diabetes Empowerment Scale Short Form (DES-SF); Likert scale; "Strongly disagree" is 1, "Somewhat disagree" is 2, "Neutral" is 3, "Somewhat Agree" is 4, and "Strongly Agree" is 5. Scores are summed and the average is taken; higher scores is more self-efficacy
Self Care - Realted to Diabetes as assessed by Self-Care questionnaire | [At 0 (baseline) and each visit (until the end of study) - 12 months]
  Multiple Choice. Questions about diabetes related self care, "How many hours per day do you currently devote to managing your glucose levels?"
CoYoT1 Care - Tools Questions | [At 12 months or Visit 4]
  Record keeping for tools to give to patients in transition to non-study visits (ie: Shared Decision Making tool and Tidepool)
Standard Care - Tools Questions | [At 12 months or Visit 4]
  Record keeping for tools to give to patients in transition to non-study visits (ie:Tidepool)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer K Raymond, MD, MCR, Principal Investigator — Children's Hospital Los Angeles
Locations (1):
- Children's Hospital, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Guljas R, Ahmed A, Chang K, Whitlock A. Impact of telemedicine in managing type 1 diabetes among school-age children and adolescents: an integrative review. J Pediatr Nurs. 2014 May-Jun;29(3):198-204. doi: 10.1016/j.pedn.2013.10.013. Epub 2013 Oct 31. PMID 24269308
- [Background] Wood JR, Miller KM, Maahs DM, Beck RW, DiMeglio LA, Libman IM, Quinn M, Tamborlane WV, Woerner SE; T1D Exchange Clinic Network. Most youth with type 1 diabetes in the T1D Exchange Clinic Registry do not meet American Diabetes Association or International Society for Pediatric and Adolescent Diabetes clinical guidelines. Diabetes Care. 2013 Jul;36(7):2035-7. doi: 10.2337/dc12-1959. Epub 2013 Jan 22. PMID 23340893
- [Background] Miller KM, Foster NC, Beck RW, Bergenstal RM, DuBose SN, DiMeglio LA, Maahs DM, Tamborlane WV; T1D Exchange Clinic Network. Current state of type 1 diabetes treatment in the U.S.: updated data from the T1D Exchange clinic registry. Diabetes Care. 2015 Jun;38(6):971-8. doi: 10.2337/dc15-0078. PMID 25998289
- [Background] Park MJ, Scott JT, Adams SH, Brindis CD, Irwin CE Jr. Adolescent and young adult health in the United States in the past decade: little improvement and young adults remain worse off than adolescents. J Adolesc Health. 2014 Jul;55(1):3-16. doi: 10.1016/j.jadohealth.2014.04.003. Epub 2014 May 10. PMID 24815958
- [Background] Monaghan M, Helgeson V, Wiebe D. Type 1 diabetes in young adulthood. Curr Diabetes Rev. 2015;11(4):239-50. doi: 10.2174/1573399811666150421114957. PMID 25901502
- [Background] American Diabetes Association. Economic costs of diabetes in the U.S. in 2012. Diabetes Care. 2013 Apr;36(4):1033-46. doi: 10.2337/dc12-2625. Epub 2013 Mar 6. PMID 23468086
- [Background] Li R, Barker LE, Shrestha S, Zhang P, Duru OK, Pearson-Clarke T, Gregg EW. Changes over time in high out-of-pocket health care burden in U.S. adults with diabetes, 2001-2011. Diabetes Care. 2014 Jun;37(6):1629-35. doi: 10.2337/dc13-1997. Epub 2014 Mar 25. PMID 24667459
- [Background] Naranjo D, Schwartz DD, Delamater AM. Diabetes in ethnically diverse youth: disparate burden and intervention approaches. Curr Diabetes Rev. 2015;11(4):251-60. doi: 10.2174/1573399811666150421115846. PMID 25901501
- [Background] Valenzuela JM, Seid M, Waitzfelder B, Anderson AM, Beavers DP, Dabelea DM, Dolan LM, Imperatore G, Marcovina S, Reynolds K, Yi-Frazier J, Mayer-Davis EJ; SEARCH for Diabetes in Youth Study Group. Prevalence of and disparities in barriers to care experienced by youth with type 1 diabetes. J Pediatr. 2014 Jun;164(6):1369-75.e1. doi: 10.1016/j.jpeds.2014.01.035. Epub 2014 Feb 25. PMID 24582008
- [Background] Lado JJ, Lipman TH. Racial and Ethnic Disparities in the Incidence, Treatment, and Outcomes of Youth with Type 1 Diabetes. Endocrinol Metab Clin North Am. 2016 Jun;45(2):453-61. doi: 10.1016/j.ecl.2016.01.002. Epub 2016 Apr 7. PMID 27241975
- [Background] Peek ME, Cargill A, Huang ES. Diabetes health disparities: a systematic review of health care interventions. Med Care Res Rev. 2007 Oct;64(5 Suppl):101S-56S. doi: 10.1177/1077558707305409. PMID 17881626
- [Background] Zuijdwijk CS, Cuerden M, Mahmud FH. Social determinants of health on glycemic control in pediatric type 1 diabetes. J Pediatr. 2013 Apr;162(4):730-5. doi: 10.1016/j.jpeds.2012.12.010. Epub 2013 Jan 26. PMID 23360562
- [Background] Hill KE, Gleadle JM, Pulvirenti M, McNaughton DA. The social determinants of health for people with type 1 diabetes that progress to end-stage renal disease. Health Expect. 2015 Dec;18(6):2513-21. doi: 10.1111/hex.12220. Epub 2014 Jun 17. PMID 24938493
- [Background] Peters A, Laffel L; American Diabetes Association Transitions Working Group. Diabetes care for emerging adults: recommendations for transition from pediatric to adult diabetes care systems: a position statement of the American Diabetes Association, with representation by the American College of Osteopathic Family Physicians, the American Academy of Pediatrics, the American Association of Clinical Endocrinologists, the American Osteopathic Association, the Centers for Disease Control and Prevention, Children with Diabetes, The Endocrine Society, the International Society for Pediatric and Adolescent Diabetes, Juvenile Diabetes Research Foundation International, the National Diabetes Education Program, and the Pediatric Endocrine Society (formerly Lawson Wilkins Pediatric Endocrine Society). Diabetes Care. 2011 Nov;34(11):2477-85. doi: 10.2337/dc11-1723. No abstract available. PMID 22025785
- [Background] Introduction. Diabetes Care. 2017 Jan;40(Suppl 1):S1-S2. doi: 10.2337/dc17-S001. No abstract available. PMID 27979885
- [Background] Orals. Diabetes. 2013 Jul;62(Supplement_1):A1-A98. doi: 10.2337/db13-1-387. No abstract available. PMID 23792714
- [Background] Dinesen B, Nonnecke B, Lindeman D, Toft E, Kidholm K, Jethwani K, Young HM, Spindler H, Oestergaard CU, Southard JA, Gutierrez M, Anderson N, Albert NM, Han JJ, Nesbitt T. Personalized Telehealth in the Future: A Global Research Agenda. J Med Internet Res. 2016 Mar 1;18(3):e53. doi: 10.2196/jmir.5257. PMID 26932229
- [Background] Garvey KC, Beste MG, Luff D, Atakov-Castillo A, Wolpert HA, Ritholz MD. Experiences of health care transition voiced by young adults with type 1 diabetes: a qualitative study. Adolesc Health Med Ther. 2014 Oct 20;5:191-8. doi: 10.2147/AHMT.S67943. eCollection 2014. PMID 25349485
- [Background] Dougherty JP, Lipman TH, Hyams S, Montgomery KA. Telemedicine for adolescents with type 1 diabetes. West J Nurs Res. 2014 Oct;36(9):1199-221. doi: 10.1177/0193945914528387. Epub 2014 Apr 1. PMID 24695401
- [Background] Franc S, Borot S, Ronsin O, Quesada JL, Dardari D, Fagour C, Renard E, Leguerrier AM, Vigeral C, Moreau F, Winiszewski P, Vambergue A, Mosnier-Pudar H, Kessler L, Reffet S, Guerci B, Millot L, Halimi S, Thivolet C, Benhamou PY, Penfornis A, Charpentier G, Hanaire H. Telemedicine and type 1 diabetes: is technology per se sufficient to improve glycaemic control? Diabetes Metab. 2014 Feb;40(1):61-66. doi: 10.1016/j.diabet.2013.09.001. Epub 2013 Oct 16. PMID 24139705
- [Background] Raymond JK. Models of Care for Adolescents and Young Adults with Type 1 Diabetes in Transition: Shared Medical Appointments and Telemedicine. Pediatr Ann. 2017 May 1;46(5):e193-e197. doi: 10.3928/19382359-20170425-01. PMID 28489225
- [Background] Lehmkuhl HD, Storch EA, Cammarata C, Meyer K, Rahman O, Silverstein J, Malasanos T, Geffken G. Telehealth behavior therapy for the management of type 1 diabetes in adolescents. J Diabetes Sci Technol. 2010 Jan 1;4(1):199-208. doi: 10.1177/193229681000400125. PMID 20167185
- [Background] Boogerd EA, Noordam C, Kremer JA, Prins JB, Verhaak CM. Teaming up: feasibility of an online treatment environment for adolescents with type 1 diabetes. Pediatr Diabetes. 2014 Aug;15(5):394-402. doi: 10.1111/pedi.12103. Epub 2013 Dec 18. PMID 24350732
- [Background] Harris MA, Freeman KA, Duke DC. Seeing Is Believing: Using Skype to Improve Diabetes Outcomes in Youth. Diabetes Care. 2015 Aug;38(8):1427-34. doi: 10.2337/dc14-2469. Epub 2015 Jun 1. PMID 26033508
- [Background] Heyworth L, Rozenblum R, Burgess JF Jr, Baker E, Meterko M, Prescott D, Neuwirth Z, Simon SR. Influence of shared medical appointments on patient satisfaction: a retrospective 3-year study. Ann Fam Med. 2014 Jul;12(4):324-30. doi: 10.1370/afm.1660. PMID 25024240
- [Background] Raymond JK, Berget CL, Driscoll KA, Ketchum K, Cain C, Fred Thomas JF. CoYoT1 Clinic: Innovative Telemedicine Care Model for Young Adults with Type 1 Diabetes. Diabetes Technol Ther. 2016 Jun;18(6):385-90. doi: 10.1089/dia.2015.0425. Epub 2016 May 19. PMID 27196443
- [Background] Raymond JK, Shea JJ, Berget C, Cain C, Fay-Itzkowitz E, Gilmer L, Hoops S, Owen D, Shepard D, Spiegel G, Klingensmith G. A novel approach to adolescents with type 1 diabetes: the team clinic model. Diabetes Spectr. 2015 Jan;28(1):68-71. doi: 10.2337/diaspect.28.1.68. No abstract available. PMID 25717281
- [Derived] Bisno DI, Reid MW, Pyatak EA, Flores Garcia J, Salcedo-Rodriguez E, Torres Sanchez A, Fox DS, Hiyari S, Fogel JL, Marshall I, Bachmann G, Raymond JK. Virtual Peer Groups Reduce HbA1c and Increase Continuous Glucose Monitor Use in Adolescents and Young Adults with Type 1 Diabetes. Diabetes Technol Ther. 2023 Sep;25(9):589-601. doi: 10.1089/dia.2023.0199. Epub 2023 Aug 17. PMID 37335751
- [Derived] Raymond JK, Reid MW, Fox S, Garcia JF, Miller D, Bisno D, Fogel JL, Krishnan S, Pyatak EA. Adapting home telehealth group appointment model (CoYoT1 clinic) for a low SES, publicly insured, minority young adult population with type 1 diabetes. Contemp Clin Trials. 2020 Jan;88:105896. doi: 10.1016/j.cct.2019.105896. Epub 2019 Nov 18. PMID 31751776